CLINICAL TRIAL: NCT02465684
Title: The Role of a Thigh Tourniquet in Unicondylar Knee Arthroplasty: a Randomized Controlled Trial
Brief Title: Effect of Tourniquet on UKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Medical University Linz, Austria (Unknown)
Responsible Party: Principal Investigator, Michael Liebensteiner, Michael Liebensteiner MD, PhD, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UKA-Tourniquet
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Tourniquets; Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- tourniquet (Experimental): UKA surgery with tourniquet
  Interventions: Procedure: unicondylar knee arthroplasty
- no tourniquet (Experimental): UKA without tourniquet
  Interventions: Procedure: unicondylar knee arthroplasty

INTERVENTIONS:
Procedure: unicondylar knee arthroplasty

SUMMARY:
There is obviously a lack of evidence regarding the risk-benefit ratio of a thigh tourniquet in unicondylar knee arthroplasty (UKA). This refers to many possible outcome criteria like operating time, blood loss, quality of prosthesis fixation in the bone, adverse events, radiographic result, clinical score outcome, easy of rehabilitation etc. It is not appropriate to rely on findings from the field of total knee arthroplasty.

It is the aim of the current study, to clarify the role of a thigh tourniquet during UKA with regard to component fixation quality, component positioning and sizing, clinical outcome and rehabilitation process.

Patients scheduled for routine UKA implantation due to osteoarthritis or osteonecrosis in the medial compartment will be considered for participation.

Patients are then randomized for surgery with or without tourniquet. After an anteromedial Quad-Sparing approach the UKA procedure itself is then carried out, as suggested by the manufacturer. For both groups puls lavage and meticulous drying is applied before cementing.

The following outcome parameters are assessed: 1)radiographic cement mantle thickness, 2)component position & sizing, 3)diolucencies, 4)score outcome and 5)parameters of early Rehab.

ELIGIBILITY:
Inclusion Criteria:

* waiting list for unicondylar knee arthroplasty

Exclusion Criteria:

* failed upper tibial osteotomy,
* insufficiency of the collateral or anterior cruciate ligaments,
* a fixed varus or valgus deformity (not passively correctable) above 15°,
* a flexion deformity greater than 15° and 5) rheumatoid arthritis. In addition - with regard to the scope of the current study - further exclusion criteria will be
* intake of medicinal anticoagulation prior to surgery
* liver dysfunction / coagulation dysfunction
* peripheral arterial obstructive disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
cement mantle thickness | 1 week